CLINICAL TRIAL: NCT05870306
Title: Triple Atria Extrastimuli vs Pulmonary Vein Isolation Alone in Persistent Atrial Fibrillation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Principal Investigator, Juan Fernandez-Armenta Pastor, PhD MD, Instituto de investigación e innovación biomédica de Cádiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCA-AF 1230-N-20
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Atrial fibrillation; Functional mapping; Hidden slow conduction
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 105 patients undergoing a first-time ablation procedure for AF will be consecutively enrolled and randomized on a 1:1 basis to PVI alone vs PVI plus slow conduction ablation.
  An enrollment log with all the patients included in the study, even drops out, will be collected. Data will be collected at enrollment, baseline and at three, six and 12-month follow-up visit.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI alone (Other): High-density voltage mapping using a multipolar catheter (PentaRay or OctaRay, Biosense Webster, Diamond Bar, CA, USA) will be performed during AF. PVI will be performed with the standard protocol. If needed electrical cardioversion will be performed after PVI ablation. A 10-minute waiting period after isolation of each ipsilateral PV pair was applied to assess for acute reconnections. Additional RF applications were performed if needed at reconnection sites until PVI was achieved.
  Interventions: Procedure: pulmonary vein isolation
- PVI PLUS HSC ABLATION (Experimental): After standard PVI isolation point-by point ablation targeting HSC-EGMs will be performed. HSC-EGMs with a distance less than 5 mm between them will be addressed with a single application. The ablation index will be defined based on the LA wall thickness (LAWT) at the location of the HSC-EGM: LAWT < 1mm: 300 f, LAWT 1-2 mm: 350 f, LAWT 2-3 mm: 400 f and LAWT >3 mm: 450 f. This is the experimental intervention added to pulmonary veins isolation. This intervention, in terms of risks, is superimposable to the ablation of CFAEs or rotational activity, which are stablished techniques for PsAF catheter ablation
  Interventions: Procedure: pulmonary vein isolation and targeted radiofrequency ablation

INTERVENTIONS:
Procedure: pulmonary vein isolation and targeted radiofrequency ablation — Radiofrequency will be delivered around the left atrial ostia to isolate the veins. Extra radiofrequency ablation will be performed on the targeted areas
  Arms: PVI PLUS HSC ABLATION
Procedure: pulmonary vein isolation — Radiofrequency will be delivered around the left atrial ostia to isolate the veins.
  Arms: PVI alone

SUMMARY:
The problem addressed in this proposal is related to the success rate in treating one of the most common arrhythmias in the Western population, atrial fibrillation (AF). Specifically, the success rate is particularly low in persistent atrial fibrillation, being up to 40% lower than the success rate for paroxysmal atrial fibrillation.

Atrial fibrillation is associated with increased mortality and morbidity (stroke, heart failure, dementia, etc.). The most effective treatment is electrical isolation of the pulmonary veins (PVI) by catheter ablation using radiofrequency or cryoablation of the atrial myocardial tissue. This ablation allows the elimination of the main initiators of the arrhythmia but may not address its maintainers, which play a significant role in persistent atrial fibrillation.

This project proposes a new approach in studying the atrial myocardial substrate for persistent fibrillation ablation. Until now, maintainers of the arrhythmia have been sought by conducting studies during atrial fibrillation. In this project, we will use short-coupled stimulation techniques during sinus rhythm and analyze the response of the atrial myocardium, attempting to unmask areas where the impulse propagates abnormally/slowly. These areas of the atrial muscle with hidden slow conduction (HSC) could generate short circuits that maintain atrial fibrillation. It would be expected that these areas would show fragmented electrograms in response to rapid electrical stimuli not visible in basal rhythm.

The study is divided into two sub-studies to be carried out over the 3-year project.

1. This study aims to test the feasibility of this new arrhythmic substrate characterization strategy, as well as observe differences between patients with paroxysmal and persistent AF and compare it with conventional fragmented electrogram analysis during AF.
2. The second sub-study will apply the knowledge acquired during the first phase regarding the characterization of electrograms-HSC, allowing for radiofrequency ablation procedures to be performed using a new substrate ablation technique consisting of the elimination of these electrograms and comparing the results with those patients who undergo conventional pulmonary vein ablation techniques.

The ultimate goal, from a global point of view, is to demonstrate that it is possible to improve the results of arrhythmia treatment by identifying and eliminating these electrograms-HSC.

DETAILED DESCRIPTION:
STUDY PURPOSE The aims of the current study are

* To investigate the presence, characteristics and location of complex electrograms suggestive of slow conduction zones elucidated by triple atria extrastimuli during sinus rhythm in paroxysmal and persistent Atrial Fibrillation (AF)
* Correlate atrial HSC- electrograms during sinus with continuously fractionated electrograms during AF in patients with persistent AF
* Test the hypothesis that elimination of atrial HSC-Electrograms(EGM) in addition to PVI would improve ablation outcomes in PersistentAF(PsAF) patients versus PVI alone in a randomized study.

Sub-study 1 (ANALYSIS OF HIDDEN SLOW CONDUCTION ELECTROGRAMS IN PAROXISMAL AND PERSISTENT ATRIAL FIBRILLATION. HSC-AF STUDY):

1.1. OBJETIVES HYPOTHESIS Left atrial EGM showing HSC elucidated by atria extrastimuli should be more manifest in persistent versus paroxysmal AF and should de more spatially and temporarily reproducible compared to fractionated EGM during AF STUDY OBJETIVES 1.1 Describe the method to elucidate HSC using a triple atrial extrastimuli 1.2 Analyze the characteristics and location of HSC-EGMs 1.3 Compare the presence, burden, characteristics and location of HSC-EGMs in paroxysmal versus persistent AF 1.4 Compare the presence and location of HSC-ECGs with fractionated EGM during AF

1.2. METHODS Summary of methods: 10 patients with paroxysmal AF and 10 patients with PsAF who undergoing a first-time ablation procedure for AF will be consecutively included to describe the complex electrograms (presence, distribution, number of deflections, amplitude, duration, delta of EGM width) elucidated by triple atria extrastimuli during sinus rhythm.

1.2.3 PREPROCEDURAL INTERVENTIONS The usual clinical protocol for preparation for AF ablation will be followed. This includes as complementary tests: blood tests, echocardiography and cardiac CT. CT images will be analyzed with ADAS-3TM (Galgo Medical, Barcelona, Spain) to obtain 3D wall thickness maps.

1.2.4 ELECTROPHYSIOLOGIC STUDY High-density voltage mapping using a multipolar catheter (PentaRay, Biosense Webster, Diamond Bar, CA, USA) will be performed during sinus rhythm in ParoxysmalAF(PxAF) patients. During mapping, manual points after a triple extrastimulus from LA appendage will be acquired to fill all color gaps on the LA map using Carto3 with an interpolation of 6 mm for the color threshold. Triple extrastimulus will be delivered at atrial effective refractory period (AERP)+60ms plus AERP + 60 ms plus AERP +40-20ms. Adequate endocardial contact will be confirmed by stable electrograms, the distance to the geometry surface.

In PsAF patients starting the procedure in AF, a high-density map will be acquired during AF. Visually detected Comlex Fractionated Atrial Electrograms(CFAE) will be annotated with pink dots. In this subgroup of patients (10 PsAF cases) a second map will be acquired to confirm the reproducibility of this methodology and compare the location and morphology of the complex electrograms between the two acquisitions. After this second map electrical cardioversion (≤3 external biphasic shock 200-360J) will be performed to restore sinus rhythm. During sinus rhythm two consecutive high-density maps with triple extrastimuli will be constructed as previously described.

1.2.5 RADIOFREQUENCY ABLATION The CARTO3® system (Biosense Webster, Diamond Bar, CA, USA) will be used for ablation. An open irrigated, 3.5-mm tip, ablation catheter (ThermoCool® SmartTouchTM, Biosense Webster, Diamond Bar, CA, USA) Will be used for mapping and ablation. First of all, a fast-anatomical map (FAM) of the PVs and the left atrium Will be acquired. PVI is performed by point-by-point RadioFrequency(RF) applications guided with ablation index (350-450 f) to create a RF circle around the PV ostia (nephroid shape). In case of a common ipsilateral vein ostium, the line was drawn around the trunk. Acute PVI was confirmed after first pass with the usual local method by demonstrating entry and exit block with the ablation catheter placed sequentially in each of the PVs. A 10-minute waiting period after isolation of each ipsilateral PV pair was applied to assess for acute reconnections. Additional RF applications were performed if needed at reconnection sites until PVI was achieved.

1.2.6 SUBSTRATE MAPS AND ATRIAL ELECTROGRAM ANALYSIS

Low-voltage areas will be defined as sites of 3 adjacent low voltage (<0.5 mV) points, which were <5 mm apart from each other.20

* Scar tissue < 0.05mV
* Healthy tissue > 0.5mV
* 0.05mV < Border Zone < 0.5mV EGMs with high electrical noise, or poor signal quality reducing accurate assessment of abnormal EGMs were discarded

The signals during sinus rhythm will be divided into 3 types according to their electrogram waveforms:

* Normal (sharp electrograms with <=3 positive or negative distinct peaks or electrogram duration <40 ms).21, 22
* Complex EGM during SR:
* Fractionated (with >4 positive or negative distinct peaks and electrogram duration >=40 ms). Highly fragmented with ≥5 peaks ±63 ms.
* Double potential: 2 or more separate deflections separate by an isoelectric interval.21, 22
* HSC-EGM: sites that show highly fragmented or double electrograms in response to triple extrastimuli, presenting normal or fractionated electrogram in sinus rhythm (see figure). Sites will be determined by visual analysis during electroanatomical mapping(EAM) acquisition and will be analyzed offline after the procedure. Delta of duration of the bipolar EGM (third stimulated atrial EGM duration - atrial EGM duration of the sinus beat prior to triple extrastimuli) in milliseconds will be recorded.

Electroanatomical maps acquired during AF will be used to draw automatic CFAE maps using the CFAE-CARTO® module with the nominal setting of SCI CFAE maps.

After the first descriptive part of the study, all patients who fulfill the inclusion criteria will be consecutively enrolled and randomized on a 1:1 basis to PVI alone vs PVI plus slow conduction ablation.

Sub-study 2 PULMONARY VEIN ISOLATION PLUS SLOW CONDUCTION ABLATION ELUCIDATED BY TRIPLE ATRIA EXTRASTIMULI VS PULMONARY VEIN ISOLATION ALONE IN PERSISTENT ATRIAL FIBRILLATION (HSC-AF TRIAL)

2.1 OBJETIVES

HYPOTHESIS Elimination of atrial HSC-EGM in addition to PVI would improve ablation outcomes in PsAF patients versus PVI alone

2.2 METHODS Summary of methods: 105 patients with PsAF who undergoing a first-time ablation procedure for AF and fulfill inclusion criteria will be consecutively enrolled and randomized on a 1:1 basis to PVI alone vs PVI plus HSC ablation.

2.2.1 ENDPOINTS PRIMARY ENDPOINT The primary end point of the study (efficacy) will be freedom from any atrial arrhythmia (other than isthmus dependent atrial flutter) without the use of antiarrhythmic drugs at 12 months after a single ablation procedure. Patients with AF that occur in the first 3 months after the ablation (blanking period) will be censored. Each episode that lasted >30s is regarded as a recurrence.

SECONDARY ENDPOINTS The following secondary endpoints will be considered: time to first persistent AF (more than 7 days) after blanking period (efficacy), any atrial arrhythmia (other than isthmus dependent atrial flutter) on antiarrhythmic drugs at 12 months after a single ablation procedure after blanking period (efficacy), AF burden (% time AF in 24h Holter) (efficacy), incidence of periprocedural complications (safety), procedure time (feasibility), fluoroscopy time (feasibility), number of RF applications (efficiency), RF delivery time (efficiency).

2.2.4 STUDY SIZE AND DURATION 105 patients undergoing a first-time ablation procedure for AF will be consecutively enrolled and randomized on a 1:1 basis to PVI alone vs PVI plus slow conduction ablation.

An enrollment log with all the patients included in the study, even drops out, will be collected. Data will be collected at enrollment, baseline and at three, six and 12-month follow-up visit.

2.3.1 BASELINE VISIT The baseline visit must be performed after the patient has signed the informed consent form and prior to the AF ablation procedure.

2.3.2 PREPROCEDURAL INTERVENTIONS The standard clinical protocol for preparation for AF ablation will be followed. This includes as complementary tests: blood tests, echocardiography and cardiac CT. CT images will be analyzed with ADAS-3TM (Galgo Medical, Barcelona, Spain) to obtain 3D wall thickness maps.

2.3.3 RANDOMIZATION Patients will be randomly assigned to each of the ablation procedures (PVI plus HSC ablation vs. PVI alone) on a 1:1 basis before the procedure

ABLATION PROTOCOL IN THE PVI PLUS HSC ABLATION GROUP:

Cardioversion will be delivered to restore SR (≤3 synchronized, biphasic direct current shocks (150 J, 200 J, and 200 J). High-density voltage mapping using a multipolar catheter (PentaRay or OctaRay, Biosense Webster, Diamond Bar, CA, USA) will be performed. During mapping, manual points after a triple extrastimulus from LA appendage will be acquired to fill all color gaps on the LA map using Carto3 with an interpolation of 6 mm for the color threshold. Triple extrastimulus will be delivered at atrial effective refractory period (AERP)+60ms plus AERP + 60 ms plus AERP +40-20ms. Adequate endocardial contact will be confirmed by stable electrograms, the distance to the geometry surface. The bandpass filter will be set at 30-500 Hz. HSC-EGM are represented with green dots and highly fragmented EGM with pink dots, double potentials in blue.

Then, PVI will be performed with the standard protocol, using entrance and exit block as the electrophysiological end point. An open irrigated, 3.5-mm tip, ablation catheter (ThermoCool® SmartTouchTM or QDot Micro™, Biosense Webster, Diamond Bar, CA, USA) was used for mapping and ablation. First of all, a fast-anatomical map (FAM) of the PVs and the left atrium was acquired. PVI is performed by point-by-point RF applications guided with ablation index (350-450 f) to create a RF circle around the PV ostia (nephroid shape). In case of a common ipsilateral vein ostium, the line was drawn around the trunk. Acute PVI was confirmed after first pass with the usual local method by demonstrating entry and exit block with the ablation catheter placed sequentially in each of the PVs. A 10-minute waiting period after isolation of each ipsilateral PV pair was applied to assess for acute reconnections. Additional RF applications were performed if needed at reconnection sites until PVI was achieved.

After PVI isolation point-by point ablation targeting HSC-EGMs will be performed. HSC-EGMs with a distance less than 5 mm between them will be addressed with a single application. The ablation index will be defined based on the LA wall thickness (LAWT) at the location of the HSC-EGM: LAWT < 1mm: 300 f, LAWT 1-2 mm: 350 f, LAWT 2-3 mm: 400 f and LAWT >3 mm: 450 f. This is the experimental intervention added to pulmonary veins isolation. This intervention, in terms of risks, is superimposable to the ablation of CFAEs or rotational activity, which are stablished techniques for PsAF catheter ablation.24

Substrate maps and atrial electrogram analysis will be performed as described in sub-study 1

ABLATION PROTOCOL IN THE PVI GROUP:

High-density voltage mapping using a multipolar catheter will be performed during AF. PVI will be performed with the standard protocol (previously described). If needed electrical cardioversion will be performed after PVI ablation. A 10-minute waiting period after isolation of each ipsilateral PV pair was applied to assess for acute reconnections. Additional RF applications were performed if needed at reconnection sites until PVI was achieved.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients undergoing a first-time ablation procedure for AF.
* Patients with persistent or long-lasting AF; persistent AF will be defined as a sustained episode lasting >7 days and <1 year; long-lasting persistent AF will be >1 year and <3 years
* Patients with PxAF; PxAF will be defined as a sustained episode lasting <7 days;
* Patients who must be willing and able to comply with all periablation and follow-up requirements
* Patients with AF who will accept the procedure of ablation
* Patients who signed the written informed consent for the study
* Patients who can endure the required follow-up.

Exclusion Criteria:

* Patients with left atrial size ≥55 mm (2-dimensional echocardiography, parasternal long-axis view)
* Patients with severe structural cardiac disease (severe mitral regurgitation, dilated cardiomyopathy, hypertrophy cardiomyopathy, other severe valvular heart diseases)
* Patients with the serum creatinine >3.5 mg/dL or creatinine clearance rate <30 mL/min;
* Patients with life expectancy <12 months;
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with lower burden of atrial fibrillation during follow-up comparing both arms | This outcome will be analyzed during the last 8 months of the project
  It will be assessed through a 24-hour holter monitor during follow-up the burden of atrial fibrillation in both study arms. It will be evaluated whether the elimination of HSC-EGM along with PVI will improve the outcomes in Persistent AF compared to those in which only PVI is performed.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | This outcome will be analyzed during the recruitment period, starting on the 9th month with a duration of 20 months
  The feasibility of the technique will be analyzed as the percentage of cases in which adverse events occurred that prevented the study from being carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Fernandez-Armenta, PhD MD, Principal Investigator — Instituto de investigación e innovación biomédica de Cádiz
Locations (1):
- F. para la Gestión de la Inv. Biomédica de Cádiz Ríos, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data from the procedures will be uploaded to an anonymized database and shared for publications
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This information will be available from the beginning of the recruitment, at the 9th month of the project with a duration of three years.
Access Criteria: All participants in this study will get a login and password to a centralized database

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT05870306/Prot_SAP_ICF_000.pdf